CLINICAL TRIAL: NCT06942481
Title: Girls Invest: A Mobile-Enabled Economic Empowerment Intervention for Girls to Reduce Risk for Partner Violence
Brief Title: Evaluating Girls Invest: A Mobile-Enabled Economic Empowerment Intervention for Girls to Reduce Risk for Partner Violence
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: San Diego State University (Other)
Collaborators: University of Ibadan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HS-2018-0195; D-0000009194-01 (Other Grant/Funding Number: Wellspring Philanthropic Fund)
Record Dates: First submitted 2025-04-09; First posted 2025-04-24 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Risk Factors for Intimate Partner Violence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Girls Invest (Experimental): Girls Invest is an app-based economic empowerment intervention to address social and economic factors associated with IPV among girls ages 15-19 in low-income communities in Ibadan, Nigeria.
  Interventions: Behavioral: Girls Invest
- Waitlist Control group (Placebo Comparator): Participants receive the intervention after they complete the 6 month follow-up survey
  Interventions: Behavioral: Waitlist control

INTERVENTIONS:
Behavioral: Girls Invest — The Girls Invest intervention involved: 1) app-based trainings on topics related to financial literacy, gender equity, and health and 2) financial resources/incentives supporting girls' education/career.
  Arms: Girls Invest
Behavioral: Waitlist control — Participants receive Girls Invest after they complete the 6 month follow-up survey.
  Arms: Waitlist Control group

SUMMARY:
The research aims to refine and evaluate Girls Invest, a newly developed economic empowerment intervention, to reduce economic and social risks associated with high rates of intimate partner violence (IPV) among adolescent girls in Ibadan, Nigeria. Girls Invest, initially developed and tested in the US, has been adapted for use in Nigeria via Phase I Wellspring support. Girls Invest participants complete gender equity and financial skills training modules via a mobile "app." Upon completion, each participant receives a financial resource of supporting girls' education/vocation (e.g., sewing machine, baking oven and pans, or funds to cover educational exams).

DETAILED DESCRIPTION:
Adolescent girls residing in low-income communities in Nigeria experience high rates of IPV. Economic vulnerability contributes to these high rates of IPV in two major ways: 1) Economic vulnerability increases financial reliance on male partners; IPV is common in these partnerships with males and financial reliance on males decreases girls' ability to leave abusive partnerships. 2) Economic vulnerability can intersect with gender-based constraints (e.g. low prioritization of limited household resources for girls' education) and create low expectations of educational/career opportunities, which can shift girls' priorities away from the participants future training/education and increase intentions to find a male partner and start a family - thereby, increasing girls' risk for relying financially on male partners and risk for IPV. By promoting young females' financial knowledge as well as social/economic expectations and opportunities, Girls Invest seeks to decrease economic vulnerability, reduce girls' financial reliance on male partnerships, and reduce girls' risk for IPV.

First, the investigators aim to pilot Girls Invest with 20 adolescent females ages 15-19; assessments will include quantitative app-based surveys and focus group discussions to assess initial feasibility, acceptability and fidelity of implementation. The investigators will refine Girls Invest with consultation from a community advisory board. Second, to determine preliminary efficacy, the investigators will implement a 2-armed randomized-controlled trial, randomizing 240 adolescent girls ages 15-19 to the Girls Invest intervention or a wait-list control condition.

Girls Invest expands previous work on economic interventions for reducing IPV, and also employs innovative mobile technology methodologies. The proposed research has potential for high impact, particularly given the increase in economic vulnerability as a result of COVID-19, especially among girls who were already living in poverty prior to the pandemic, as well as the coinciding reports of increased IPV.

ELIGIBILITY:
Inclusion Criteria:

* Girls ages 15-19 in selected secondary classes of 16 schools in Ibadan

Exclusion Criteria:

* Girls under 15 and over 19 years of age
* Do not attend one of the selected secondary classes of 16 schools in Ibadan

Ages: 15 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — girls
Enrollment: 240 (Actual)
Dates: Start 2022-09-07 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Attitudes supportive of traditional gender roles: Gender Equitable Men (GEM) Scale | baseline to 6 months follow up
  seven items adapted from Gender Equitable Men (GEM) Scale assessing male and female roles in the following: decision-making (e.g., when to have sex, household purchases), household chores, childcare, reproductive decisions (including pregnancy prevention), and in receiving education/training. Responses involved 5-point Likert scales ranging from strongly agree to strongly disagree.
Attitudes supportive of IPV: Items adapted from Demographic Health Surveys | baseline to 6 months follow up
  7 validated items adapted from Demographic Health Surveys asking whether any of the following scenarios a husband has good reason to hit his wife: (1) She does not complete housework to his satisfaction, (2) She disobeys him, (3) She refuses to have sexual relations with him, (4) She asks him whether he has other girlfriends, (5) He finds out she has been unfaithful, (6) She goes out without telling him, or (7) She does not prepare a meal to his satisfaction. Responses involved 5-point Likert scales ranging from strongly agree to strongly disagree.
Coping with experiences of gender-based discrimination | baseline to 6 months follow up
  three items assessing perceived ability to identify instances of "gender-based discrimination against me" and coping with such experiences as being able to "take care of myself," and recognizing that such experiences are not "about anything I did as an individual; items developed based on previous literature on the topic and investigator's previous research, given the absence of a validated scale. Measure was piloted with 5 participants and refined prior to implementation.
Perceptions of economic vulnerability | baseline to 6 months follow up
  eight items asking about perceived household economic situation, including having enough money to purchase basic necessities (e.g., food, clothes, other needs) and money to pay for education/training of the participant. Items also assessed perceived financial stress of the household. Responses involved 5-point Likert scales ranging from strongly agree to strongly disagree. Scale was developed based on investigator's research and existing literature on this topic, given the lack of a validated scale. It was piloted among 5 participants prior to implementation.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Reed, Principal Investigator — San Diego State University; Olufunmilayo Fawole, Principal Investigator — University of Ibadan
Locations (1):
- University of Ibadan, Ibadan, Nigeria

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-04-23): https://cdn.clinicaltrials.gov/large-docs/81/NCT06942481/Prot_SAP_000.pdf